CLINICAL TRIAL: NCT04242342
Title: Phase II of Adaptative Magnetic Resonance-Guided Stereotactic Body Radiotherapy (SBRT) for Treatment of Primary or Secondary Progressive Liver Tumors
Brief Title: Adaptative MR-Guided Stereotactic Body Radiotherapy of Liver Tumors
Acronym: RASTAF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RASTAF IRM
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Radiotherapy
Keywords: liver cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patient with a localized primary tumor (hepatocellular carcinoma or cholangiocarcinoma) or a secondary hepatic localization of a solid carcinoma, with one to three hepatic lesions accessible to a treatment by stereotactic radiotherapy.
  Interventions: Radiation: Adaptative MR-Guided Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Adaptative MR-Guided Stereotactic Body Radiotherapy — If lesion near organs at risk:
  * Prescription of 50 Gy in 5 fractions of 10 Gy
  * 3 sessions per week, with MRI guided stereotactic radiotherapy and daily adaptive treatment
  If lesion far of organs at risk:
  * Prescription of 60 Gy in 6 fractions of 10 Gy
  * 3 sessions per week, with MRI guided stereotactic radiotherapy without daily adaptive treatment

SUMMARY:
Hepatic metastases are common in solid cancers (up to 30% of patients with colorectal cancer and up to 50% of patients during their follow-up). The incidence of primary liver cancer increases due to the increase in chronic liver diseases induced by excessive alcohol consumption, hepatitis B and C viruses, and excess fat in the liver. Surgical excision of these liver lesions is the reference treatment but it cannot always be realised.

Stereotactic radiotherapy is a recent technique proposed to hepatic metastases treatment from solid cancers and primary hepatic lesions (HCC or cholangiocarcinomas); it is possible to deliver high doses of radiation in the most conformational way possible in order to limit the irradiation of the non-tumor liver. The results of this stereotactic radiotherapy are currently very good with control rates of 75 to 80% at 1 and 2 years with acceptable rates of severe toxicities of 10%. However, the fear of hepatic, digestive (colon, esophagus, stomach) or even cardiac toxicities limits its using to the majority of patients because coupled with a conventional scanner it do not allow direct visualization of the lesion.

Due to its non-irradiating nature, MRI guided stereotactic radiotherapy can generate continuous imaging, during the irradiation session, offering " in live " a visualization of the tumor target and organs at risk of proximity. In increasing the precision and safety in the delivery of irradiation, it allows to hope for several areas for improvement of treatment:

* reduced uncertainty margins
* an increase in the dose delivered
* the accessibility of tumor lesions near sensitive organs (esophagus, stomach, heart chambers, intestines, duodenum, right kidney).

More, this accelerator allows a re-optimization of the initial dosimetric plan to the anatomical changes of the day to allow an MRI guided adaptive radiotherapy.

DETAILED DESCRIPTION:
The MRI guided stereotactic radiotherapy of hepatic lesions with an MRIdian® Linac tested in this study will allow:

* to see the tumor target in live with a non-irradiating imaging
* a reduction of the volume of non-tumor liver irradiated at high doses
* An progession of the dose delivered to the tumor lesion to allow tumor control to be increased.
* a new dosimetric plan adapted each day to the new contours to avoid a risk of severe digestive toxicity while ensuring optimal treatment, at an appropriate dose, of the tumor volume.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman aged 18 or over.
2. Performance Status 0 or 1.
3. Primary or secondary liver tumor(s)
4. maximum 1 to 3 liver tumor(s) accessible to stereotaxic body radiotherapy therapy.
5. ASAT and ALAT <3 times the upper limit of normal,
6. Albuminemia ≥ 28g / L.
7. Creatinine clearance> 30ml / min
8. signing of informed consent.
9. Woman of childbearing age who accepts effective contraception during the course of treatment and within 3 months of treatment.
10. Patient affiliated to a social security scheme.

Exclusion Criteria:

1. MRI contraindication
2. Pregnant or breastfeeding woman.
3. Patient with decompensated liver cirrhosis or cirrhosis> Child B7
4. Patient previously irradiated in the planned treatment area.
5. Refusal of patient's consent.
6. Patient unable to give his consent, under guardianship or unable to submit to the treatment protocol or protocol follow-up.
7. History of another malignant tumor except:

   * Malignant neoplasm treated with curative intent and with no known active disease ≥ 5 years before inclusion,
   * Non-melanoma or malignant lentigo skin cancer treated adequately without signs of disease,
   * Carcinoma in situ treated without sign of disease,
   * Prostate carcinoma that did not require curative treatment.
8. Known hypersensitivity to gadolinium or other gadolinium chelates.
9. Patient participating in another therapeutic trial which would require the administration of experimental treatment during the period between inclusion and the end of radiotherapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2029-01-20 (Estimated); Study Completion 2029-01-20 (Estimated)

PRIMARY OUTCOMES:
local control at 2 years | 2 years
  lack of progression according to RECIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc, Dijon, France